CLINICAL TRIAL: NCT00933972
Title: Effect of Renal Impairment on Pharmacodynamics and Pharmacokinetics of RO4998452: A Multiple-center, Open-label, Parallel Group Study Following Single Oral Dosing of RO4998452 to Type 2 Diabetes Patients With Varying Degrees of Renal Impairment.
Brief Title: A Study of RO4998452 in Type 2 Diabetes Patients With Varying Degrees of Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP22321; 2008-008128-34
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (4):
- 1 (normal) (Experimental)
  Interventions: Drug: RO4998452
- 2 (mild) (Experimental)
  Interventions: Drug: RO4998452
- 3 (moderate) (Experimental)
  Interventions: Drug: RO4998452
- 4 (severe) (Experimental)
  Interventions: Drug: RO4998452

INTERVENTIONS:
Drug: RO4998452 — 20mg po single dose

SUMMARY:
This 4 arm study will investigate the pharmacodynamics and pharmacokinetics of RO4998452 in type 2 diabetes patients with varying degrees of renal impairment. Eligible patients will be divided into 4 groups, with normal renal function, or mild, moderate or severe renal impairment. All patients will receive a single oral dose of RO4998452 in the fasted state.The anticipated time on study treatment is <3 months (single dose study)and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 40-80 years of age;
* type 2 diabetes;
* normal renal function, or impaired but stable renal function;
* stable with regard to medication or treatment regimen taken for renal impairment or diabetes.

Exclusion Criteria:

* patients with a renal transplant;
* end-stage renal disease, requiring dialysis;
* nephrotic syndrome, or a history of nephrectomy;
* type 1 diabetes mellitus.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Creatinine clearance; Pk parameters; adverse events | Days 1-3

SECONDARY OUTCOMES:
Blood glucose; meal tolerance test | Days 1-3

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Renton, Washington, United States
- Moscow, Russia